CLINICAL TRIAL: NCT04420195
Title: Pilot Study Comparing Early Conversion to Extended-Release Tacrolimus (ENVARSUS XR) to Immediate-Release Tacrolimus in Lung Transplant Recipients
Brief Title: Envarsus XR in Lung Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-01247
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Lung Transplant
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Envarsus XR (Experimental): Envarsus XR to be initiated once patient is tolerating oral medications
  Interventions: Drug: Extended-Release Tacrolimus
- IR tacrolimus (historical control) (Experimental): Historical cohort of patients maintained on IR tacrolimus following transplant
  Interventions: Drug: Immediate-Release Tacrolimus

INTERVENTIONS:
Drug: Extended-Release Tacrolimus — Envarsus XR is an FDA-approved drug for the prophylaxis of organ rejection in de novo kidney transplant patients or in kidney transplant patients converted from IR tacrolimus when used with other immunosuppressants. Envarsus XR is a novel extended-release formulation of tacrolimus created using MeltDose technology. Envarsus XR is available in tablet form. It is available in 0.75, 1, and 4 mg tablets.
  Other Names: Envarsus XR
  Arms: Envarsus XR
Drug: Immediate-Release Tacrolimus — Historical cohort of 20 subjects who will be maintained on IR tacrolimus following transplant. Dosing will be converted on an individual basis (Capsules: 0.5 mg, 1 mg and 5 mg or Injection: 5 mg) . All patients will be initiated on IR tacrolimus either under the tongue (sublingual) or as a solution given through a tube placed through the nose into the stomach, which is standard of care for all lung transplant recipients.
  Other Names: Prograf
  Arms: IR tacrolimus (historical control)

SUMMARY:
Patients undergoing a lung transplant will be enrolled. All patients will undergo lung transplantation with standard post-operative management, including triple immunosuppression. As soon as the patient is deemed appropriate to take medications via the oral route, they will be converted from IR tacrolimus to Envarsus XR. Patients will be followed per site's standard of care.

DETAILED DESCRIPTION:
Lung transplantation will be performed per standard-of-care techniques. All post-transplant management, including initial triple immunosuppression, will be carried out per standard of care. Once the patient is able to take medications via the oral route, they will be converted to Envarsus XR, which will be maintained for the first year post-lung transplant.

ELIGIBILITY:
Inclusion Criteria:

Prospective arm:

* Age ≥ 18 years
* Received a lung transplant at NYU Langone Health
* Be able to convert to Envarsus XR within the first month post-transplant
* Able and willing to provide informed consent

Historical control:

* Age ≥ 18 years
* Received a lung transplant at NYU Langone Health
* Completed one year from transplant on IR tacrolimus

Exclusion Criteria:

Prospective arm:

* Contraindication to tacrolimus due to allergic or adverse reactions
* Pregnant or nursing women
* Multi-organ transplant recipient

Historical control:

* Contraindication to tacrolimus due to allergic or adverse reactions (not including chronic kidney disease)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Angel, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD collected for this study will be used for the sole purpose of this study.

REFERENCES:
- [Derived] Lewis TC, Hotchkis P, Wong A, Lamaina V, Fitzpatrick E, Stiefel A, Ohanian J, Schnier JR, Lesko M, Rudym D, Natalini JG, Angel LF. Comparison of Early Conversion to LCP-Tacrolimus (ENVARSUS XR) to Immediate-Release Tacrolimus in Lung Transplant Recipients. Clin Transplant. 2025 May;39(5):e70159. doi: 10.1111/ctr.70159. PMID 40294109

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 41 individuals were enrolled to participate in the trial; 1 individual did not begin treatment in the study, thus, only 40 participants started the study. Data on 24 historical control individuals were collected and analyzed retrospectively for the secondary outcome measures, but these 24 individuals were not recruited nor enrolled into the study, thus, they are not reflected in the total Protocol Enrollment figure.
Groups:
- IR Tacrolimus (Historical Control): Historical cohort of patients maintained on IR tacrolimus following transplant. These patients were not enrolled in the trial as participants.
  Immediate-Release Tacrolimus: Historical cohort of 20 subjects who will be maintained on IR tacrolimus following transplant. Dosing will be converted on an individual basis (Capsules: 0.5 mg, 1 mg and 5 mg or Injection: 5 mg) . All patients will be initiated on IR tacrolimus either under the tongue (sublingual) or as a solution given through a tube placed through the nose into the stomach, which is standard of care for all lung transplant recipients.
Period: Overall Study
Arm/Group | Envarsus XR | IR Tacrolimus (Historical Control)
Started | 40 | 24
Completed | 40 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Envarsus XR | IR Tacrolimus (Historical Control) | Total
Number analyzed (Participants) | 40 | 24 | 64
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 59 [47 to 66] | 62.5 [56 to 68] | 60.75 [47 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 25 | 16 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 7 | 25
  Not Hispanic or Latino | 22 | 17 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 18 | 7 | 25
Region of Enrollment [Number; unit: participants]
  United States | 40 | 24 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Remaining on Envarsus XR at 1 Year
Description: The primary endpoint is the percentage of patients remaining on Envarsus XR at the 1-year follow-up visit.
Time Frame: 1 Year Post-Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Envarsus XR
Number analyzed (Participants) | 40
Participants | 40

2. Secondary Outcome: Freedom From Acute Cellular Rejection (ACR) at 1 Year
Description: Number of participants who did not experience ACR as of the 1-year follow-up.
Time Frame: Up to 1 Year Post-Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Envarsus XR | IR Tacrolimus (Historical Control)
Number analyzed (Participants) | 40 | 24
Participants | 5 | 6

3. Secondary Outcome: Composite Rejection Standardized Score (CRSS)
Description: The CRSS is a novel measure of burden of ACR. The score ranges from 0-6; higher scores indicate greater severity of burden of ACR.
Time Frame: 1 Year Post-Transplant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Envarsus XR | IR Tacrolimus (Historical Control)
Number analyzed (Participants) | 40 | 24
score on a scale | 0.19 (0.37) | 0.33 (0.43)

4. Secondary Outcome: Number of Treated Episodes of ACR
Description: Number of participants with treated episodes of biopsy-proven or clinically suspected rejection requiring treatment with intravenous methylprednisolone or anti-thymocyte globulin.
Time Frame: Up to 1 Year Post-Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Envarsus XR | IR Tacrolimus (Historical Control)
Number analyzed (Participants) | 40 | 24
Participants | 8 | 6

5. Secondary Outcome: Number of Participants With of Chronic Lung Allograft Dysfunction (CLAD)
Description: Number of participants with at least 1 instance of CLAD.
Time Frame: Up to 1 Year Post-Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Envarsus XR | IR Tacrolimus (Historical Control)
Number analyzed (Participants) | 40 | 24
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With De Novo Donor-Specific Antibody (DSA)
Description: Number of individuals in whom an antibody is detected after transplantation.
Time Frame: Up to 1 Year Post-Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Envarsus XR | IR Tacrolimus (Historical Control)
Number analyzed (Participants) | 40 | 24
Participants | 19 | 4

7. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR)
Description: Change in Estimated Glomerular Filtration Rate (eGFR) at 1 year post-transplant from pre-transplant.
Time Frame: Baseline, 1 Year Post-Transplant
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Envarsus XR | IR Tacrolimus (Historical Control)
Number analyzed (Participants) | 40 | 24
mL/min/1.73m2 | -56.2 (27.1) | -40.3 (21.2)

8. Secondary Outcome: Overall Survival at 1 Year
Description: The percentage of participants who are alive at 1 year post-transplant.
Time Frame: 1 Year Post-Transplant
Measure: Number; unit: Percentage of participants
Arm/Group | Envarsus XR | IR Tacrolimus (Historical Control)
Number analyzed (Participants) | 40 | 24
Percentage of participants | 100 | 100

ADVERSE EVENTS:
Time Frame: 2 years.
Description: Adverse events were assessed through regular investigator assessment and laboratory testing in the Envarsus XR group only. Adverse event data (adverse event/serious adverse events) were not collected from/assessed in the Historical Control group. All-cause mortality was assessed in both groups, via the outcome measure "Overall Survival."
Groups:
- Historical Controls: Historical cohort of patients maintained on IR tacrolimus following transplant. These patients were not enrolled in the trial as participants.
  Immediate-Release Tacrolimus: Historical cohort of 20 subjects who will be maintained on IR tacrolimus following transplant. Dosing will be converted on an individual basis (Capsules: 0.5 mg, 1 mg and 5 mg or Injection: 5 mg) . All patients will be initiated on IR tacrolimus either under the tongue (sublingual) or as a solution given through a tube placed through the nose into the stomach, which is standard of care for all lung transplant recipients.
Arm/Group | Envarsus XR | Historical Controls
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/0
Other Adverse Events (participants affected / at risk) | 29/40 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Envarsus XR (N=40) | Historical Controls (N=0)
Allograft failure (Injury, poisoning and procedural complications) | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Envarsus XR (N=40) | Historical Controls (N=0)
Sepsis/pneumonia (Infections and infestations) | 8 | NA
Acute rejection (Injury, poisoning and procedural complications) | 9 | NA
Nausea/vomiting/diarrhea (Gastrointestinal disorders) | 7 | NA
Respiratory viral infection (Infections and infestations) | 5 | NA
Hyperglycemia/Hyperosmolar hyperglycemic state (HHS)/Diabetic ketoacidosis (DKA) (Metabolism and nutrition disorders) | 3 | NA
Hyponatremia (Metabolism and nutrition disorders) | 2 | NA
Video-assisted thoracoscopic surgery (VATS) pleurodesis (Surgical and medical procedures) | 2 | NA
Cytomegalovirus (CMV) infection (Infections and infestations) | 2 | NA
Antibody-mediated rejection (Injury, poisoning and procedural complications) | 2 | NA
Pleural effusion/thoracentesis (Respiratory, thoracic and mediastinal disorders) | 2 | NA
Diverticulitis (Gastrointestinal disorders) | 2 | NA
Anxiety attack (Psychiatric disorders) | 1 | NA
Mycobacterium avium-intracellulare (MAI) infection (Infections and infestations) | 1 | NA
Peripheral neuropathy/pain (Nervous system disorders) | 1 | NA
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Sinusitis (Infections and infestations) | 1 | NA
Ureterostomy (Renal and urinary disorders) | 1 | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Dysphagia/aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Hypotension/syncope (Vascular disorders) | 1 | NA
Pericarditis (Cardiac disorders) | 1 | NA
Drug overdose (Injury, poisoning and procedural complications) | 1 | NA
Arrhythmia (Cardiac disorders) | 1 | NA
Aspergillus infection (Infections and infestations) | 1 | NA
Acute kidney injury (Renal and urinary disorders) | 1 | NA
Hemoptysis after transbronchial biopsy (Injury, poisoning and procedural complications) | 1 | NA
Cough/shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT04420195/Prot_SAP_000.pdf